CLINICAL TRIAL: NCT00965341
Title: A Preliminary Trial of Testosterone Replacement for Fatigue in Male Hypogonadic Patients With Advanced Cancer.
Brief Title: Testosterone Replacement for Fatigue in Male Hypogonadic Advanced Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008-0262
Record Dates: First submitted 2009-08-21; First posted 2009-08-25 (Estimated); Results first posted 2016-09-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-07

CONDITIONS: Advanced Cancer
Keywords: Cancer; Fatigue; Testosterone Replacement Therapy; Depo-Testosterone; Testosterone cypionate; Testosterone enanthate; Hypogonadic; Functional Assessment of Cancer Therapy-Fatigue subscale; FACIT-F
MeSH Terms: conditions — Neoplasms; Fatigue | interventions — Testosterone; testosterone enanthate; testosterone 17 beta-cypionate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Testosterone (Active Comparator): Testosterone Starting dose of 150 or 200 mg testosterone enanthate/cypionate by injection into buttock muscle, every 15 days through Day 72.
  Interventions: Drug: Testosterone
- Placebo (Placebo Comparator): Starting dose of 150 mg or 200 mg sesame seed oil by injection into buttock muscle, about every 15 days through Day 72.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Testosterone — Starting dose of 150 or 200 mg testosterone enanthate/cypionate by injection into buttock muscle, every 15 days through Day 72.
  Other Names: Androderm; AndroGel; Delatestryl; Depo-Testosterone; Testosterone enanthate; Testosterone cypionate
  Arms: Testosterone
Drug: Placebo — Starting dose of 150 mg or 200 mg sesame seed oil by injection into buttock muscle, about every 15 days through Day 72.
  Arms: Placebo

SUMMARY:
The goal of this clinical research study is to learn if and how testosterone replacement therapy may affect fatigue in males with advanced cancer and low testosterone levels.

DETAILED DESCRIPTION:
Background for Study:

Testosterone is the main sex hormone for males. Cancer, cancer treatments and cancer symptoms can cause its levels in the body to drop below normal. When testosterone is taken as a drug (called "testosterone replacement therapy"), this therapy is designed to return the testosterone levels to normal. This may help to control symptoms of low testosterone levels, which may include fatigue.

In addition to fatigue, low testosterone levels may also cause depression, loss of sexual desire, loss of appetite, and/or physical changes such as effects on strength, stamina (long-lasting strength and energy), energy level, and body composition. In this study, researchers also want to learn how testosterone therapy may affect these other symptoms that may occur. To measure these effects, questionnaires and other tests will be used.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups. One group will receive testosterone, and the other group will receive a placebo. A placebo is a substance that looks like the study drug but has no active ingredients. There is an equal chance that you will be assigned to either group.

Neither you, the study doctor, nor the study staff will know whether you are receiving testosterone or placebo until Day 72. However, if needed for your safety, the study doctor and staff will be able to find out which one you are receiving.

You will receive testosterone or placebo by injection into your buttock muscle, about every 15 days until Day 72 (+/- 3 days). This is at baseline (+/- 3 days), Day 15 (+/- 3 days), Day 29 (+/- 3 days), Day 43 (+/- 3 days), and Day 57 (+/- 3 days).

As part of the routine blood tests performed at your study visits, your testosterone levels will be measured. If your testosterone level is too high, your testosterone/placebo dose will be lowered. If your testosterone level is too low, your testosterone/placebo dose will be raised.

Baseline Visit:

On Day 1, you will have a series of tests performed.

Your strength and stamina will be measured by hand-grip strength tests, a Get-Up-and-Go test and a 6-minute walk test.

* For the hand-grip strength tests, you will grip a device with your hand as hard as you can. You will repeat both of these tests 3 times for each hand.
* For the Get-Up-and-Go test, you will be timed to see how long it takes you to get up from sitting in a chair, walk 10 feet, turn around and walk back to the chair, and sit down.
* For the 6-minute walk test, you will be timed while you walk on a 100-foot loop. You will walk 50 feet and then turn and walk back to the beginning. You will do this at a walking speed that feels comfortable and for as many times as you can in 6 minutes.

A muscle on your upper arm will be measured. This will be the arm you do not normally use for writing.

You will be weighed on a scale that measures your body composition. Body composition includes measurements of your body fat, "lean" (non-fat) body weight, and how much water is in your body.

Blood (about 1-2 tablespoons) will be drawn for research on inflammation, other proteins and hormones. These tests are designed to help researchers learn if testosterone affects inflammation and/or fatigue, and if increased levels of certain hormones may help increase muscle and appetite.

You will be given a device called an Actiwatch, which is worn like a wristwatch. It will measure your physical activity. The research staff will show you how to use it. You should wear it through Day 29 of the study. You will return it at your Day 15 and Day 29 study visit.

Other Study Visits:

On Days 15, 29, 43, 57 and 72 (all +/- 3 days), the following tests and procedures will be performed:

* Blood (about 1 tablespoon) will be drawn for routine tests.
* You will complete questionnaires.
* Your strength and stamina, arm muscle, and body composition will be measured.
* A medical history and physical exam will be performed on Day 29 (+/-3 days) and Day 72 (+/3 days)

If your questionnaire responses show that you may be having emotional difficulties or depression, you will be provided with names of mental health providers in case you would like to receive mental health screening.

Length of Study:

You may remain on study until Day 72. You will be taken off study early if intolerable side effects occur, the cancer gets worse, or the fatigue gets worse.

Optional Open-Label Testosterone Dosing:

At your Day 72 visit, you will find out if you were receiving testosterone or placebo. Those participants who were receiving testosterone will be given the option to keep receiving testosterone (off-study). Those participants who were receiving the placebo will also be given the option to receive testosterone (off-study). This is called "Open-Label Testosterone Dosing."

If you choose to receive testosterone off-study after Day 72, you will receive testosterone by injection into your buttock muscle.

This is an investigational study. Testosterone replacement therapy is commercially available and FDA approved for use in men with HIV, for treating low testosterone levels and fatigue. (HIV is a virus that affects the immune system.) At this time, it is investigational to use testosterone replacement therapy to treat low testosterone levels and fatigue in patients with cancer.

Up to 126 patients will take part in this multicenter study. Up to 80 patients will be enrolled at M. D. Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients with any advanced cancer (metastatic or locally recurrent) who have a bioavailable testosterone (BT) of < 70 ng/dL.
2. Male patients who have fatigue present every day for the last two weeks and have an Edmonton Symptom Assessment System (ESAS) fatigue score during the last 24 hours of >/= to 4 on a 0 to 10 scale (in which 0 = no fatigue and 10 = worst possible fatigue).
3. Male patients who are willing to receive intramuscular injections every 2 weeks and are 18 years of age or older are eligible for this study.
4. Participants must be willing to have blood samples drawn at screening and/or baseline and every two weeks until the end of treatment.
5. Prostatic Specific Antigen (PSA) level must be lower than 4.0 ng/mL to be eligible for this study and Digital Rectal Exam (DRE) must be normal.
6. Eastern Cooperative Oncology Group (ECOG) PS </= 3 and participants must be able to stand up with or without assistance and to ambulate.
7. Hemoglobin (Hgb) >/= 9 g/dL. If the patient has not had blood drawn for a hemoglobin level in the past 28 days, one will be done to determine eligibility. Patients with a hemoglobin < 9 g/dL will be referred for treatment of their anemia.

Exclusion Criteria:

1. Patients who are determined incapable of completing questionnaires due to cognitive or physical deficits are ineligible for this study
2. Abnormal Digital Rectal Exam (DRE) at baseline or history of severe untreated benign prostatic hypertrophy (BPH) with International Prostatic Symptom Score (IPSS) >19.
3. Patients with a history of prostate cancer, a history of breast cancer or adenocarcinoma of unknown origin.
4. A history of untreated obstructive sleep apnea.
5. Uncontrolled severe heart failure (NYHA Class III or IV), uncontrolled cardiac arrhythmia or severe chronic obstructive pulmonary disease (COPD) requiring home oxygen.
6. Patients who have evidence of pre-existing hypopituitarism/hypogonadism including status post bilateral orchiectomy, for which replacement therapy is mandated, are ineligible for this study.
7. Patients exhibiting clinically diagnosed severe dehydration are ineligible.
8. Patients with a history of uncontrolled arrhythmia.
9. Patients who are currently receiving androgen therapy or dehydroepiandrosterone (DHEA)
10. Diabetics with a history of frequent episodes of hypoglycemia or uncontrolled diabetes mellitus (DM) defined as a fasting glucose over 200 mg/dL or HbA1c above 8%.
11. Uncontrolled thyroid disease
12. Hypercalcemia (corrected calcium > 10.5 g/dL); estimated glomerular filtration rate < 60 mg/min using the Modification of Diet in Renal Disease glomerular filtration rate (MDRD GFR); ALT > 3x the upper limit of normal (UNL)
13. Patients on warfarin, cyclosporine, dong quai, eucalyptus, dicumarol, germander, Jin bu huan, kava, pennyroyal, chaparral, comfrey, phenprocoumon are ineligible for this study.
14. Unstable symptoms could contribute to fatigue such as severe pain (score> 6 on ESAS) or severe depression (defined as a score of 15 or greater on the Depression Subscale of the Hospital Anxiety Depression Scale [HADS]). These symptoms should be resolved or stable for >/= 2 weeks at baseline for inclusion into study.
15. Patients with hematocrit (Hct) > upper normal limits (UNL) will be excluded due to possible polycythemia. If the patient has not had blood drawn for a hematocrit level in the past 28 days, one will be performed at baseline to determine eligibility.
16. Patients who have a known sensitivity to sesame seed products.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2009-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rony Dev, DO, Principal Investigator — UT MD Anderson Cancer Center
Locations (2):
- United States (2):
  - The DeBakey VA Medical Center/Baylor College of Medicine, Houston, Texas
  - UT MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinic outpatients with advanced cancer were recruited from September 2009 to November 2011 at both Michael E. DeBakey Veterans Affairs Medical Center (VA) and University of Texas MD Anderson Cancer Center (MDACC).
Pre-assignment Details: Of the 53 participants enrolled only 43 subjects met eligibility criteria. Ten participants either did not meet criteria or withdrew consent prior to assignment to groups.
Period: Overall Study
Arm/Group | Testosterone | Placebo
Started | 19 | 24
Completed | 13 | 16
Not Completed | 6 | 8
Not completed — Withdrew consent | 1 | 5
Not completed — Lost to Follow-up | 1 | 0
Not completed — Transportation issues | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Testosterone | Placebo | Total
Number analyzed (Participants) | 19 | 24 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 7 | 13 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 19 | 24 | 43
Region of Enrollment [Number; unit: participants]
  United States | 19 | 24 | 43

OUTCOME MEASURES:

1. Primary Outcome: Functional Assessment of Cancer Therapy-Fatigue Subscale (FACIT-F) at Day 29 (+/- 3 Days)
Description: The primary endpoint was to evaluate the effect of testosterone replacement therapy on fatigue in hypogonadic male patients with advanced cancer, measured by the Functional Assessment of Cancer Therapy-Fatigue subscale (FACIT-F) at day 29 (+/- 3 days). FACIT-F consists of 27 general quality-of-life questions divided into 4 domains (physical, social, emotional, and functional), plus a 13-item fatigue subscore. The participant rates the intensity of fatigue and its related symptoms on a scale of 0-4. The FACIT-F total score ranged between 0 and 108, with higher scores denoting improved function. The FACIT-F Fatigue Subscale ranges from 0 to 52, with higher scores represent better (less) fatigue than a lower score. A positive difference score (29 days minus baseline) represents improvement. A greater positive difference score represents greater improvement.
Time Frame: Day 29 (+/- 3 days)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 13 | 16
units on a scale
  FACIT-F Total Score (29 days-baseline) | 12 (13.8) | 13 (19.3)
  FACIT-F Fatigue Subscale (29 days-baseline) | 12 (7.7) | 14 (12.0)

2. Secondary Outcome: The Hospital Anxiety and Depression Scale (HADS) and Symptoms Scored by the Edmonton Symptom Assessment Scale (ESAS).
Description: The ESAS assessed 10 symptoms experienced by cancer patients during the previous 24 hours: pain, fatigue, nausea, depression, anxiety, drowsiness, dyspnea, anorexia, sleep disturbance, and feelings of well-being. The severity of each symptom is rated on a numerical scale of 0-10 (0 = no symptom, 10 = worst possible severity). Depression was assessed using the 14-item HADS questionnaire. Each item on the questionnaire was scored from 0-3. Total Scores for the HADS Questionnaire range from 0 to 42 with higher scores denoting feeling of depression.
Time Frame: Day 29 (+/- 3 days)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 13 | 16
units on a scale
  Anxiety, ESAS | 7 (3) | 5 (2)
  Depression, HADS | 7 (3) | 6 (3)
  Well being, ESAS | 5 (3) | 3 (3)
  Sleep, ESAS | 5 (2) | 4 (2)
  Appetite, ESAS | 5 (3) | 4 (3)
  Dyspnea, ESAS | 2 (3) | 3 (2)
  Drowsiness, ESAS | 5 (3) | 4 (2)
  Nausea, ESAS | 2 (2) | 2 (3)
  Fatigue, ESAS | 6 (2) | 6 (2)
  Pain, ESAS | 3 (2) | 3 (2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline through day 57 and 30 days after the last study drug injection.
Arm/Group | Testosterone | Placebo
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/24
Other Adverse Events (participants affected / at risk) | 13/19 | 9/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone (N=19) | Placebo (N=24)
Death (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone (N=19) | Placebo (N=24)
Fatigue (General disorders) | 2 (2) | 3 (3)
Pain (NOS) (General disorders) | 2 (2) | 1 (1)
Anorexia (General disorders) | 2 (2) | 2 (2)
Dyspnea (General disorders) | 0 (0) | 3 (3)
Neuropathy: Sensory (General disorders) | 2 (2) | 0 (0)
Hemoglobin (General disorders) | 1 (1) | 0 (0)
Infection (Other) (General disorders) | 1 (1) | 0 (0)
Neuropathy: Cranial (General disorders) | 1 (1) | 0 (0)
Pain (Other) (General disorders) | 1 (1) | 0 (0)
Pain (Skin) (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study has several limitations; the follow-up visits at two weekly intervals were burdensome for many patients. Others did not want to enroll in a placebo-controlled trial, and many patients regarded the intramuscular injections as too painful.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No